CLINICAL TRIAL: NCT01292304
Title: Single Center, Open Labeled Pilot Study Evaluating the Safety and Efficacy of Tolvaptan in Patients With Cirrhotic Ascites
Brief Title: Tolvaptan for Ascites in Cirrhotic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-IST-10-06
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Ascites; Cirrhosis
Keywords: Cirrhotic; Tolvaptan; v2 receptor antagonist
MeSH Terms: conditions — Ascites; Fibrosis | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan (Experimental): Tolvaptan 15 mg tablet once daily for 7 days followed by Tolvaptan 30 mg (two 15 mg tablets) once daily according to efficacy and tolerability
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Oral administration once daily Dosage will range from 15 mg to 30 mg
  Other Names: (SAMSCA)

SUMMARY:
Open Label Study evaluating the safety and efficacy of tolvaptan in the treatment of ascites in liver cirrhosis. Tolvaptan will be administered in combination with current ascites management.

DETAILED DESCRIPTION:
This is an open label, 12 week dose escalating pilot study of tolvaptan (initiating at 15 mg a day and increasing to 30 mg a day as tolerated in addition to standard ascites treatment) of 10 cirrhotic subjects meeting all inclusion/exclusion criteria. Subjects are monitored for changes in frequency of paracentesis, quantity of ascites removed, and body weight. Additionally, subjects laboratory values were checked frequently during the first days of dosing to ensure tolerability and slow correction/increase in serum sodium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of liver confirmed by histology and/or combination of ultrasound or endoscopic examination with laboratory evidence
* Clinically evident ascites treated by diet and/or diuretics
* History of 1 or more therapeutic paracentesis in the previous 6 months.

Exclusion Criteria:

* History of variceal bleeding
* Current or history of Gastrointestinal bleeding within 10 days of screening
* Ascites from another cause other than liver cirrhosis (i.e. cardiac origin, peritoneal infection, or peritoneal carcinoma)
* INR (International normalized ratio) > 3.0, neutrophils <1500 cell/μl, platelets < 40,000/μl
* serum bilirubin > 3 mg/dl
* serum sodium < 125 meQ (milliequivalent)/L
* serum potassium <3.5 meQ/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe (Joseph) Morelli, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Hepatology, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tolvaptan
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 62.5 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worsening Ascites (Increase in Number of Paracentesis Procedures to Remove 2 Liters of Ascites Fluid)
Description: Increase in number of therapeutic paracentesis (removal of > 2 litres of ascites fluid) during 12 weeks of study drug dosing versus 12 weeks before study drug dosing
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Number of Patients With Reduction of Ascites (Weight Loss of 2 kg or More)
Description: Number of patients with reduction of ascites is defined as reduction of weight by at least 2 kg during study drug dosing
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
participants | 0

3. Secondary Outcome: Number of Patients With Abnormally Low Levels of Sodium (Sodium Levels Between 130 mmol/L and 135 mmol/L)
Description: Number of Patients with new episodes of hyponatremia (abnormally low levels of sodium) defined as sodium >130 mmol/L and <135 mmol/L
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
participants | 1

4. Primary Outcome: Number of Subjects With Worsening Ascites (Defined as Greater Than 2 kg Weight Gain)
Description: This outcome will provide the number of subjects with a weight increase of > 2kg from baseline (worsening ascites)
Time Frame: 12 weeks of study drug
Measure: Number; unit: participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
participants | 7

5. Secondary Outcome: Time From Baseline to Worsening Ascites (Requiring 1 or More Therapeutic Paracentesis to Remove Ascites Fluid)
Description: This outcome will describe the average time from baseline for subjects to require a therapeutic paracentesis to remove ascites fluid.
Time Frame: 12 weeks of study drug
Measure: Median (Full Range); unit: Days
Arm/Group | Tolvaptan
Number analyzed (Participants) | 10
Days | 27 [8 to 57]

ADVERSE EVENTS:
Time Frame: Adverse events collected from baseline day 1 of study drug through day 99 (2 weeks after last dose)
Arm/Group | Tolvaptan
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=10)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Asterixis (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Cold Sensitivity (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Dry mouth (General disorders) | 2 (2)
Elevated serum creatinine (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyopmagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hypernatrimia (Blood and lymphatic system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (2)
Lethargy (General disorders) | 1 (1)
Lung pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth soreness (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Nighttime blackouts (Nervous system disorders) | 1 (1)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polydipsia (General disorders) | 8 (8)
Polyphagia (Metabolism and nutrition disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No